CLINICAL TRIAL: NCT04035122
Title: Effects of Robotic Neurorehabilitation With Lokomat on Physiological Responses in Neurological Patients: a Randomized Controlled Trial
Brief Title: Physiological Responses in Robotic Neurorehabilitation
Acronym: Lokophysio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Medical Director, Neurologist, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRCCSME:15/2019
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Interventional Study
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study is a parallel-group randomized clinical trial using a double-blind study design. The enrolled patients will be randomly assigned to the 2 groups using an automated computerized randomization program. Patients will be informed about the research and will be asked to fill in the informed consent form. The patient's basic characteristics (age, sex, duration of the illness, marital status and educational background) will be recorded. Randomization will be performed using a randomization list, so patients will be randomized in a 1:1 ratio in the intervention or control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list is blind to anyone involved in informing potential study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Treatment (Experimental): The Lokomat is a robotic device. For treatment with the robotic system, the amount of body weight supported will initially set at 70% of every patient's weight, then decreasing in accordance with load tolerance, although not providing less than 20% support. The selected speed will be adapted to the patient's working comfort under the supervision of a trained physiotherapist. The rehabilitation protocol consists of 40 training sessions (3 sessions per week lasting 45 minutes).
  Interventions: Other: Robotic Treatment
- Conventional Treatment (Active Comparator): The CG will perform traditional overgroung gait rehabilitation. Exercises in this program are designed with gradual increments to meet each patient's abilities and were supervised by a physical therapist. The rehabilitation protocol consists of 40 training sessions (3 sessions per week lasting 45 minutes).
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Robotic Treatment — The Lokomat is a robotic device, consisting of a powered gait orthosis with integrated computer-controlled linear actuators at each hip and knee joint, a body weight support, and a treadmill. During the Lokomat training, the patients completed at least 30 min of treatment session.
  Other Names: Lokomatdevice
  Arms: Robotic Treatment
Other: Conventional Treatment — The standard physical treatment program consisted of general conditioning exercises, including warming up (e.g. calf, shoulder, and hand passive range of motion exercises), lower and upper extremity strengthening, postural control exercises. During the conventional training, the patients completed at least 30 min of treatment session.
  Other Names: control group
  Arms: Conventional Treatment

SUMMARY:
Robotic rehabilitation is very useful for improving functional recovery in neurological patients, there is not much evidence on its role in improving physiological responses (i.e. intestinal motility, orthostatic pressure), which are often abnormal in these patients.

To this end, we designed a randomized controlled experimental study on neurological patients, with the aim of evaluating the effects of robotic neurorehabilitation using Lokomat on physiological responses, compared to traditional therapy.

ELIGIBILITY:
Inclusion criteria: diagnosis of neurological disease; age between 18 and 75; and Caucasian ethnicity; a FIM motor score equal to or greater than 30.

Exclusion criteria: patients with a history of concomitant brain surgery; severe cognitive or language impairment; systemic, bone or joint disorders; presence of disabling sensory alterations; concomitant medical and psychiatric illness that could interfere with VR training.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Constipation Scoring System | 8 months
  Constipation Scoring System (CSS) is an eight-element self-report measure designed to assess the prevalence and severity of constipation. The authors used a pathophysiological definition of constipation. The scoring system is based on eight variables (frequency of bowel movements; difficult or painful evacuation; completeness of evacuation; abdominal pain; time per attempt; assistance including laxatives; digits or enemas; number of failed evacuation attempts in a period of 24 hours and duration of constipation). The CSS consists of seven objects that are marked using a five-point Likert scale ranging from 0 (no time) to 4 (all the time) and an article evaluated on a 0-2 scale. A total score can range from 0 (normal) to 30 (severe constipation). A limit score of 15 suggests constipation.
Delta of variation in maximum and minimum blood pressure | 8 months
  Orthostatic pressure derives from systolic pressure and / or diastolic blood pressure (BP) (about 10 mm / Hg) from supine to vertical. It is evaluated by delta of variation in maximum and minimum blood pressure.

SECONDARY OUTCOMES:
The 12-Item Short Form Health Survey | 8 months
  The SF-12 Health Survey (SF-12) is a 12-article questionnaire used to assess general health outcomes from a patient's perspective. SF-12 assesses health-related quality of life, including the impact of all diseases on a wide range of functional domains. SF-12 consists of a subset of 12 articles dealing with physical functioning, physical role, physical pain, general health, vitality, social functioning, emotional role and mental health.
Functional Independence Measure | 8 months
  The FIM scale is a questionnaire that evaluates 18 activities of daily life (13 motor-sphincteric, 5 cognitive). Each activity can receive a variable score between 1 (complete dependence on others) and 7 (complete self-sufficiency). The cumulative score and the profile of the scores in the different items represent standard indicators that are now very common in the world of rehabilitation. The applications range from the measurement of the appropriateness and effectiveness of the rehabilitation intervention on the individual case, to the forecast of hospitalization times, care interviews and health costs in single operational units or on the network, or in longitudinal "path" rehabilitation studies. The cumulative scores produce a quantitative index of the person's disability.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco S Calabrò, MD, Principal Investigator — IRCCS Centro Neurolesi
Locations (1):
- IRCCS Neurolesi, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calabro RS, Russo M, Naro A, De Luca R, Leo A, Tomasello P, Molonia F, Dattola V, Bramanti A, Bramanti P. Robotic gait training in multiple sclerosis rehabilitation: Can virtual reality make the difference? Findings from a randomized controlled trial. J Neurol Sci. 2017 Jun 15;377:25-30. doi: 10.1016/j.jns.2017.03.047. Epub 2017 Mar 29. PMID 28477702
- [Result] Calabro RS, Cacciola A, Berte F, Manuli A, Leo A, Bramanti A, Naro A, Milardi D, Bramanti P. Robotic gait rehabilitation and substitution devices in neurological disorders: where are we now? Neurol Sci. 2016 Apr;37(4):503-14. doi: 10.1007/s10072-016-2474-4. Epub 2016 Jan 18. PMID 26781943